CLINICAL TRIAL: NCT00967005
Title: N-Acetyl Cysteine Plus Behavioral Therapy for Nicotine Dependent Pathological Gamblers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0908M70981; 1RC1DA028279-01 (NIH)
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-02

CONDITIONS: Gambling; Tobacco Use Disorder
Keywords: N acetyl cysteine; Pathological gambling; Nicotine dependence
MeSH Terms: conditions — Gambling; Tobacco Use Disorder | interventions — Acetylcysteine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N Acetyl Cysteine (Experimental): The objective of this application is to examine whether, given its mechanism of action, the dietary supplement, N-acetyl cysteine (NAC) will reduce both tobacco use and PG symptoms in nicotine dependent pathological gamblers.
  Interventions: Drug: N Acetyl Cysteine
- Sugar Pill (Placebo Comparator)
  Interventions: Other: Sugar Pill

INTERVENTIONS:
Drug: N Acetyl Cysteine — N-Acetyl Cysteine, 1200mg-3000mg each day for 24-weeks
  Other Names: N-acetylcysteine, Acetylcysteine, NAC
  Arms: N Acetyl Cysteine
Other: Sugar Pill — placebo control
  Arms: Sugar Pill

SUMMARY:
The objective of this application is to examine whether, given its mechanism of action, the dietary supplement, N-acetyl cysteine (NAC) will reduce both tobacco use and pathological gamblers (PG) symptoms in nicotine dependent pathological gamblers.

DETAILED DESCRIPTION:
Among US adults, 12.8% report nicotine dependence, and nicotine dependence is highly associated with a variety of DSM-IV Axis I and II disorders (Grant BF et al., 2004). Pathological gambling (PG), a serious public health problem with detrimental effects on individuals and families, and with an estimated yearly cost to society of 5 billion dollars due to lost jobs, debt, bankruptcy, and incarcerations, is associated with elevated proportions of nicotine dependence (41% - 55%), and tobacco smoking in clinical samples of pathological gamblers has been associated with increased gambling severity and more frequent psychiatric problems (Smart & Ferris, 1996; Crockfod & El-Guebaly, 1998; Shaffer et al., 1999; Petry & Oncken, 2002; Potenza et al., 2004; Grant et al., 2005; Falk et al., 2006; Fagan et al., 2007). In addition, research suggests that continued nicotine use is associated with greater rates of relapse among pathological gamblers who received behavioral therapy. Despite increased awareness of the relationship between nicotine dependence and PG, and the possible effects of nicotine dependence on gambling severity, no previous research has focused on how assessment and treatment of nicotine dependence may aid in the successful treatment of PG or smoking cessation. Preliminary research suggests that behavioral therapy using imaginal desensitization and motivational interviewing (IDMI) has shown promise in reducing the symptoms of PG (Grant et al., in press). Despite the efficacy of treatments for PG and nicotine dependence, relapse is common among individuals with nicotine dependence and PG. Preclinical studies have suggested that levels of glutamate within the nucleus accumbens mediate reward-seeking behavior and may underlie relapse seen in addictions. N-acetyl cysteine, a dietary supplement, amino acid and cysteine pro-drug, appears to modulate glutamate within the nucleus accumbens and has shown benefit in reducing the reward-seeking behavior in individuals with cocaine dependence and in pathological gamblers (Baker et al., 2003; LaRowe et al., 2006; Grant et al., 2006). If successful in treating nicotine dependent pathological gamblers, N-acetyl cysteine may serve as a viable, low-cost, and easily available treatment option for nicotine dependent pathological gamblers who receive behavioral therapy.

We therefore propose to examine how a dietary supplement, N-acetyl cysteine, used in combination with behavioral therapy, will affect both the urge to smoke and gamble in nicotine dependent pathological gamblers and smoking and gambling behaviors. We therefore propose a randomized placebo-controlled trial of N-acetyl cysteine or placebo with 80 nicotine dependent pathological gamblers who will all receive brief standardized smoking cessation treatment (Ask, Advise, and Refer model) for nicotine cessation and 6 sessions of IDMI for PG. We hypothesize that N-acetyl cysteine plus behavioral therapy will result in greater reduction in both nicotine dependence and PG symptoms during the acute treatment phase and will enhance greater long-term abstinence. Our research will contribute to an improved understanding of the treatment of nicotine-dependent pathological gamblers as well as a greater understanding of the treatment of co-occurring addictions. If our intervention is successful, it will have the potential to set a new standard of care for a range of psychiatric disorders that co-occur with nicotine dependence.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients, age 18-75 years;
2. Presence of current DSM-IV nicotine dependence and PG for at least 6 months duration;
3. Stable psychotropic drug dose for a period of at least 3 months prior to study entry;
4. Completion of complete blood count, urinalysis, liver function tests, thyroid function tests, and pregnancy test with no evidence of significant lab abnormalities;
5. Signed informed consent

Exclusion Criteria:

1. Subjects who are currently receiving individual or group therapy specifically for nicotine dependence or PG symptoms;
2. Currently receiving pharmacotherapies for either nicotine dependence or pathological gambling;
3. Subjects who have started attending Gamblers Anonymous within the 3 months prior to study initiation;
4. Subjects who have an unstable and significant medical illness;
5. Current clinically significant suicidality (score or 3 or 4 on item 3 of the Hamilton Depression Rating Scale) or any other disorder requiring immediate intervention;
6. Lifetime history of bipolar disorder type I or II, dementia, or psychotic disorder;
7. Current (past 12 months) DSM-IV substance abuse or dependence (except nicotine dependence);
8. Borderline or antisocial personality disorder based on the SCID-II;
9. Positive urine drug screen at screening;
10. Asthma (given possible worsening of asthma due to NAC);
11. Cognitive impairment that interferes with the capacity to understand and self-administer medication or provide written informed consent;
12. Current pregnancy or lactation, or inadequate contraception in women of childbearing potential; and
13. Previous treatment with NAC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc N Potenza, MD, PhD, Principal Investigator — Yale University; Jon E Grant, MD, JD, MPH, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Minnesota School of Medicine, Minneapolis, Minnesota

REFERENCES:
- [Derived] Dowling N, Merkouris S, Lubman D, Thomas S, Bowden-Jones H, Cowlishaw S. Pharmacological interventions for the treatment of disordered and problem gambling. Cochrane Database Syst Rev. 2022 Sep 22;9(9):CD008936. doi: 10.1002/14651858.CD008936.pub2. PMID 36130734
- [Derived] Grant JE, Odlaug BL, Chamberlain SR, Potenza MN, Schreiber LR, Donahue CB, Kim SW. A randomized, placebo-controlled trial of N-acetylcysteine plus imaginal desensitization for nicotine-dependent pathological gamblers. J Clin Psychiatry. 2014 Jan;75(1):39-45. doi: 10.4088/JCP.13m08411. PMID 24345329
- [Derived] Potenza MN, Balodis IM, Franco CA, Bullock S, Xu J, Chung T, Grant JE. Neurobiological considerations in understanding behavioral treatments for pathological gambling. Psychol Addict Behav. 2013 Jun;27(2):380-92. doi: 10.1037/a0032389. Epub 2013 Apr 15. PMID 23586456

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N Acetyl Cysteine | Sugar Pill
Started | 13 | 15
Treatment Completion | 10 | 10
Completed | 6 | 5
Not Completed | 7 | 10
Not completed — Lost to Follow-up | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N Acetyl Cysteine | Sugar Pill | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (10.1) | 47.7 (10.6) | 47.6 (10.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 15 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Yale-Brown Obsessive Compulsive Scale Modified for Pathological Gambling Total Score
Description: Week 0 corresponds to baseline. Minimum score=0 and maximum score=40, with higher score signifying more severe symptoms. Scale is 10 items scored from 0 to 4. Scores on each item are summed to compute total score. Thoughts/urges (questions 1 to 5) and behavior (questions 6 to 10) are added to get the total score.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 23.5 (6.4) | 20.4 (5.0)

2. Primary Outcome: Yale-Brown Obsessive Compulsive Scale Modified for Pathological Gambling Total Score
Description: Week 6 corresponds to end of N-acetylcysteine plus Ask-Advise-Refer therapy versus placebo plus Ask-Advise-Refer therapy. Minimum score=0 and maximum score=40, with higher score signifying more severe symptoms. Scale is 10 items scored from 0 to 4. Scores on each item are summed to compute total score. Thoughts/urges (questions 1 to 5) and behavior (questions 6 to 10) are added to get the total score.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 17.4 (9.1) | 16.3 (7.4)

3. Primary Outcome: Yale-Brown Obsessive Compulsive Scale Modified for Pathological Gambling Total Score
Description: Week 12 corresponds to end of 6 sessions of N-acetylcysteine plus imaginal desensitization and motivational interviewing versus placebo plus imaginal desensitization and motivational interviewing. Minimum score=0 and maximum score=40, with higher score signifying more severe symptoms. Scale is 10 items scored from 0 to 4. Scores on each item are summed to compute total score. Thoughts/urges (questions 1 to 5) and behavior (questions 6 to 10) are added to get the total score.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 7.5 (4.6) | 5.5 (5.9)

4. Primary Outcome: Yale-Brown Obsessive Compulsive Scale Modified for Pathological Gambling Total Score
Description: Week 24 represents the 3-month follow-up period (ie, corresponds to being off N-acetylcysteine or placebo and done with imaginal desensitization and motivational interviewing for 12 weeks). Minimum score=0 and maximum score=40, with higher score signifying more severe symptoms. Scale is 10 items scored from 0 to 4. Scores on each item are summed to compute total score. Thoughts/urges (questions 1 to 5) and behavior (questions 6 to 10) are added to get the total score.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 1.0 (1.3) | 6.4 (6.2)

5. Primary Outcome: Yale-Brown Obsessive Compulsive Scale Modified for Pathological Gambling Urges/Thoughts Subscale
Description: Week 0 corresponds to baseline. Questions 1 through 5 are summed to compute the thoughts/urges subscale. Minimum=0 and maximum=20, with higher scores signifying more severe thoughts/urges.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 11.8 (3.7) | 9.0 (3.4)

6. Primary Outcome: Yale-Brown Obsessive Compulsive Scale Modified for Pathological Gambling Urges/Thoughts Subscale
Description: Week 6 corresponds to end of N-acetylcysteine plus Ask-Advise-Refer therapy versus placebo plus Ask-Advise-Refer therapy. Questions 1 through 5 are summed to compute the thoughts/urges subscale. Minimum=0 and maximum=20, with higher scores signifying more severe thoughts/urges.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 8.9 (4.2) | 7.9 (3.8)

7. Primary Outcome: Yale-Brown Obsessive Compulsive Scale Modified for Pathological Gambling Urges/Thoughts Subscale
Description: Week 12 corresponds to end of 6 sessions of N-acetylcysteine plus imaginal desensitization and motivational interviewing versus placebo plus imaginal desensitization and motivational interviewing. Questions 1 through 5 are summed to compute the thoughts/urges subscale. Minimum=0 and maximum=20, with higher scores signifying more severe thoughts/urges.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 5.5 (2.3) | 2.7 (2.1)

8. Primary Outcome: Yale-Brown Obsessive Compulsive Scale Modified for Pathological Gambling Urges/Thoughts Subscale
Description: Week 24 represents the 3-month follow-up period (ie, corresponds to being off N-acetylcysteine or placebo and done with imaginal desensitization and motivational interviewing for 12 weeks). Questions 1 through 5 are summed to compute the thoughts/urges subscale. Minimum=0 and maximum=20, with higher scores signifying more severe thoughts/urges.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 0.8 (1.2) | 3.6 (3.6)

9. Primary Outcome: Yale-Brown Obsessive Compulsive Scale Modified for Pathological Gambling Behavior Subscale
Description: Week 0 corresponds to baseline. Questions 6 through 10 are summed to compute the thoughts/urges subscale. Minimum=0 and maximum=20, with higher scores signifying more severe gambling behaviors.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 11.7 (3.7) | 11.4 (2.8)

10. Primary Outcome: Yale-Brown Obsessive Compulsive Scale Modified for Pathological Gambling Behavior Subscale
Description: Week 6 corresponds to end of N-acetylcysteine plus Ask-Advise-Refer therapy versus placebo plus Ask-Advise-Refer therapy. . Questions 6 through 10 are summed to compute the thoughts/urges subscale. Minimum=0 and maximum=20, with higher scores signifying more severe gambling behaviors.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 8.5 (5.7) | 8.3 (4.9)

11. Primary Outcome: Yale-Brown Obsessive Compulsive Scale Modified for Pathological Gambling Behavior Subscale
Description: Week 12 corresponds to end of 6 sessions of N-acetylcysteine plus imaginal desensitization and motivational interviewing versus placebo plus imaginal desensitization and motivational interviewing. Questions 6 through 10 are summed to compute the thoughts/urges subscale. Minimum=0 and maximum=20, with higher scores signifying more severe gambling behaviors.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 2.0 (3.1) | 2.8 (4.5)

12. Primary Outcome: Yale-Brown Obsessive Compulsive Scale Modified for Pathological Gambling Behavior Subscale
Description: Week 24 represents the 3-month follow-up period (ie, corresponds to being off N-acetylcysteine or placebo and done with imaginal desensitization and motivational interviewing for 12 weeks). Questions 6 through 10 are summed to compute the thoughts/urges subscale. Minimum=0 and maximum=20, with higher scores signifying more severe gambling behaviors.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 0.2 (0.4) | 2.8 (4.1)

13. Primary Outcome: Fagerstrom Test for Nicotine Dependence Total Score
Description: Week 0 corresponds to baseline. This scale has 6 questions. Questions 1 and 4 are on a scale from 0 to 3 (higher scores being more severe symptoms) and questions 2, 3, 5, and 6 are on a scale from 0 to 1 (1 being more severe symptoms). Scores on all questions are summed to compute total score, with higher total score meaning more severe nicotine dependence. Scores range from 0 to 10.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 6.5 (2.0) | 6.7 (2.1)

14. Primary Outcome: Fagerstrom Test for Nicotine Dependence Total Score
Description: Week 6 corresponds to end of N-acetylcysteine plus Ask-Advise-Refer therapy versus placebo plus Ask-Advise-Refer therapy. This scale has 6 questions. Questions 1 and 4 are on a scale from 0 to 3 (higher scores being more severe symptoms) and questions 2, 3, 5, and 6 are on a scale from 0 to 1 (1 being more severe symptoms). Scores on all questions are summed to compute total score, with higher total score meaning more severe nicotine dependence. Scores range from 0 to 10.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 4.0 (1.9) | 5.9 (2.4)

15. Primary Outcome: Fagerstrom Test for Nicotine Dependence Total Score
Description: Week 12 corresponds to end of 6 sessions of N-acetylcysteine plus imaginal desensitization and motivational interviewing versus placebo plus imaginal desensitization and motivational interviewing. This scale has 6 questions. Questions 1 and 4 are on a scale from 0 to 3 (higher scores being more severe symptoms) and questions 2, 3, 5, and 6 are on a scale from 0 to 1 (1 being more severe symptoms). Scores on all questions are summed to compute total score, with higher total score meaning more severe nicotine dependence. Scores range from 0 to 10.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 5.3 (2.9) | 5.0 (1.5)

16. Primary Outcome: Fagerstrom Test for Nicotine Dependence Total Score
Description: Week 24 represents the 3-month follow-up period (ie, corresponds to being off N-acetylcysteine or placebo and done with imaginal desensitization and motivational interviewing for 12 weeks). This scale has 6 questions. Questions 1 and 4 are on a scale from 0 to 3 (higher scores being more severe symptoms) and questions 2, 3, 5, and 6 are on a scale from 0 to 1 (1 being more severe symptoms). Scores on all questions are summed to compute total score, with higher total score meaning more severe nicotine dependence. Scores range from 0 to 10.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 4.6 (1.3) | 5.3 (1.2)

17. Primary Outcome: Hamilton Depression Rating Scale Total Score
Description: Week 0 corresponds to baseline. This scale assesses depressed mood, feelings of guilt, difficulty sleeping, somatic symptoms, and others. Total score is computed by summing the scores of the 17 items. Minimum score is 0 and maximum score is 52, with higher scores signifying more severe depressive symptoms.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 9.7 (5.7) | 7.9 (4.8)

18. Primary Outcome: Hamilton Depression Rating Scale Total Score
Description: Week 6 corresponds to end of N-acetylcysteine plus Ask-Advise-Refer therapy versus placebo plus Ask-Advise-Refer therapy. This scale assesses depressed mood, feelings of guilt, difficulty sleeping, somatic symptoms, and others. Total score is computed by summing the scores of the 17 items. Minimum score is 0 and maximum score is 52, with higher scores signifying more severe depressive symptoms.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 7.5 (4.7) | 5.5 (3.8)

19. Primary Outcome: Hamilton Depression Rating Scale Total Score
Description: Week 12 corresponds to end of 6 sessions of N-acetylcysteine plus imaginal desensitization and motivational interviewing versus placebo plus imaginal desensitization and motivational interviewing. This scale assesses depressed mood, feelings of guilt, difficulty sleeping, somatic symptoms, and others. Total score is computed by summing the scores of the 17 items. Minimum score is 0 and maximum score is 52, with higher scores signifying more severe depressive symptoms.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 7.0 (4.9) | 3.7 (3.2)

20. Primary Outcome: Hamilton Depression Rating Scale Total Score
Description: Week 24 represents the 3-month follow-up period (ie, corresponds to being off N-acetylcysteine or placebo and done with imaginal desensitization and motivational interviewing for 12 weeks). This scale assesses depressed mood, feelings of guilt, difficulty sleeping, somatic symptoms, and others. Total score is computed by summing the scores of the 17 items. Minimum score is 0 and maximum score is 52, with higher scores signifying more severe depressive symptoms.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 2.8 (2.1) | 3.5 (1.7)

21. Primary Outcome: Hamilton Anxiety Rating Scale Total Score
Description: Week 0 corresponds to baseline. This scale measures anxiety symptoms, tension, somatic symptoms, difficulty concentrating, and others. Total score is computed by summing the scores on the 14 items (each item is scored from 0 to 4). Minimum score= 0 and maximum score= 56, with higher scores signifying more severe anxiety symptoms.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 11.1 (10.8) | 9.7 (6.6)

22. Primary Outcome: Hamilton Anxiety Rating Scale Total Score
Description: Week 6 corresponds to end of N-acetylcysteine plus Ask-Advise-Refer therapy versus placebo plus Ask-Advise-Refer therapy. This scale measures anxiety symptoms, tension, somatic symptoms, difficulty concentrating, and others. Total score is computed by summing the scores on the 14 items (each item is scored from 0 to 4). Minimum score= 0 and maximum score= 56, with higher scores signifying more severe anxiety symptoms.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 7.5 (4.3) | 6.2 (4.0)

23. Primary Outcome: Hamilton Anxiety Rating Scale Total Score
Description: Week 12 corresponds to end of 6 sessions of N-acetylcysteine plus imaginal desensitization and motivational interviewing versus placebo plus imaginal desensitization and motivational interviewing. This scale measures anxiety symptoms, tension, somatic symptoms, difficulty concentrating, and others. Total score is computed by summing the scores on the 14 items (each item is scored from 0 to 4). Minimum score= 0 and maximum score= 56, with higher scores signifying more severe anxiety symptoms.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 7.4 (3.2) | 4.2 (3.2)

24. Primary Outcome: Hamilton Anxiety Rating Scale Total Score
Description: Week 24 represents the 3-month follow-up period (ie, corresponds to being off N-acetylcysteine or placebo and done with imaginal desensitization and motivational interviewing for 12 weeks). This scale measures anxiety symptoms, tension, somatic symptoms, difficulty concentrating, and others. Total score is computed by summing the scores on the 14 items (each item is scored from 0 to 4). Minimum score= 0 and maximum score= 56, with higher scores signifying more severe anxiety symptoms.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 13 | 15
units on a scale | 5.0 (3.6) | 6.5 (5.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire 12 weeks each of the subjects were enrolled in the study.
Arm/Group | N Acetyl Cysteine | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No